CLINICAL TRIAL: NCT01509573
Title: Family-Based Prevention of Mental Health Problems in HIV/AIDS-Affected Children (R34MH084679-01A1)
Brief Title: Pilot Feasibility Trial of the Family Strengthening Intervention in Rwanda (FSI-R)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Partners in Health (Other); Harvard University (Other); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Theresa Betancourt, Associate Professor of Child Health and Human Rights, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RPCGA-FSI-15440
Record Dates: First submitted 2011-12-22; First posted 2012-01-13 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Depressive Symptoms; Anxiety; Parenting
Keywords: prevention therapy; depressive symptoms; anxiety; parenting; family functioning; resilience, psychological; Developing countries; Rwanda; HIV/AIDS
MeSH Terms: conditions — Depression; Anxiety Disorders; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FSI-R (Intervention group) (Experimental): The intervention group will participate in the mental health assessments and FSI-R, and will participate in post-intervention assessments and follow-up assessments.
  Interventions: Behavioral: Family Strengthening Intervention in Rwanda (FSI-R)
- TAU (Treatment as Usual) (No Intervention): The TAU control group will not receive any intervention, but will participate in treatment as usual as provided by Partners In Health. They will complete assessments at all three time points.

INTERVENTIONS:
Behavioral: Family Strengthening Intervention in Rwanda (FSI-R) — Core components of the FSI-R are derived from the FBPI theoretical framework, and were chosen to address key risk factors identified in qualitative data. The FSI-R holds separate preliminary meetings with caregivers and children to prepare for a larger family meeting. In these modules, the interventionist helps caregivers and children prioritize concerns or key messages that they most want to share with the other party. Role play and discussions are used to impart improved parenting and communication skills. In the family meetings, children and caregivers share their concerns with one another and develop a shared family narrative, which integrates past events into a singular story with shared goals and a future orientation. These family modules also discuss the services and supports (formal and non-formal resources) that the family can engage with in order to achieve their shared goals.
  8-12 weeks for 1-2 hours per week, depending on each family's pace and coverage of the material.
  Arms: FSI-R (Intervention group)

SUMMARY:
The research will examine the following Specific Aims:

Specific Aim 1: To adapt a U.S.-developed family-focused and strengths-based prevention program to the context of HIV/AIDS-affected families in Rwanda (the Family-Strengthening Intervention in Rwanda or "FSI-R") using prior qualitative findings and CAB input.

Specific Aim 2: To deliver the intervention to a small group of families to collect preliminary data on intervention feasibility, acceptability, and to further refine the intervention manual for the FSI-R.

Specific Aim 3: To conduct a pilot feasibility study of the FSI-R with 80 families.

In pursuit of Specific Aim 3, this research will (a) conduct a preliminary exploratory analysis to examine the extent to which the FSI-R for HIV/AIDS-affected families is associated with improved caregiver-child relationships using measures of family connectedness, good parenting, and social support. Hypothesis 1: Participants in the FSI-R will demonstrate increases in protective processes compared to usual care controls not exposed to the FSI-R. It will also (b) conduct a preliminary exploratory analysis to determine the extent to which improved caregiver-child relationships are sustained four months after the conclusion of the FSI-R. Hypothesis 2: Four months after the conclusion of the intervention, participants in the FSI-R will demonstrate increases in protective processes compared to usual care controls not exposed to the FSI-R.

DETAILED DESCRIPTION:
The challenge of this project is to develop a family-based intervention to prevent mental health problems in children affected by HIV/AIDS that can be initiated as caregivers come into contact with health systems via routine HIV testing and care. Specifically, we propose to develop and pilot test a prevention-oriented family-strengthening intervention to mitigate the mental health risks facing HIV/AIDS-affected children (i.e., those who are HIV+ themselves or who have an HIV+ family member, including those who have died). The intervention design, which is based upon the Family-Based Preventive Intervention (FBPI), is centrally focused on galvanizing mechanisms of resilience in children and families and building on local sources of strength. Our unique adaptation and pilot study will employ a family focus to attend to the reality that HIV/AIDS is a family disease, and to show that individual, familial, and community resources may help families to succeed despite chronic illness. The pilot intervention will use a randomized design, drawing study participants (N=80 families) from social work referrals. Protective factors characterizing the family and mental health problems in children and caregivers will be assessed pre- and post-intervention. In addition, we will survey both participants and interventionists to provide qualitative and quantitative data on the program's cultural acceptability and feasibility, and on their own satisfaction.

ELIGIBILITY:
Inclusion criteria: All participants must be HIV/AIDS-affected (i.e., having an HIV+ family member, including those who have died). We will select single and dual caregiver families to reflect population dynamics in the area. Caregivers must be at least 18 years of age (the age of majority in Rwanda), must live in the same household as the children, and must be the child's legal guardian. Legal guardians may be aunts, uncles, grandparents, or foster parents. Caregivers must be willing to discuss HIV/AIDS with school-aged children in the family.

Exclusion Criteria: Potential participants will be excluded if they do not live in the Rwinkwavu catchment area. Untreated mental illness or active suicidal ideation/attempts in the family also constitutes exclusion criteria (mental health treatment for these problems may occur in conjunction with the FSI). HIV-positive children are ineligible for the study if their HIV status has not been disclosed to them. Exclusion criteria also include lack of caregiver willingness to discuss HIV/AIDS with school-aged children in the family. Youth-headed households will be excluded due to concerns about youth caregivers' capacity to participate in the FSI in addition to other caretaking duties.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Mental Health of Children and Caregivers | Administered to caregivers and school-aged children in each cohort three times: once within 15 days prior to the start of the intervention, once within 15 days of intervention completion, and again 4 months following intervention completion.
  The Mental Health Assessment Batteries for Children and Caregivers are comprehensive surveys addressing a range of locally-relevant mental health problems and protective processes, as well as issues like functioning, stigma, hope, harsh parenting, parent-child relationships, and other risk and protective factors. The mental health components of the assessments have been subject to a validation study in this community. They were developed using qualitative data gathered from this population in 2007 and 2009.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa S Betancourt, ScD, MA, Principal Investigator — Associate Professor, Harvard School of Public Health
Locations (1):
- Partners In Health/Inshuti Mu Buzima (PIH/IMB), Rwinkwavu, Rwanda

REFERENCES:
- [Background] Beardslee WR. Prevention and the clinical encounter. Am J Orthopsychiatry. 1998 Oct;68(4):521-33. doi: 10.1037/h0080361. PMID 9809112
- [Background] Beardslee WR, Gladstone TR, Wright EJ, Cooper AB. A family-based approach to the prevention of depressive symptoms in children at risk: evidence of parental and child change. Pediatrics. 2003 Aug;112(2):e119-31. doi: 10.1542/peds.112.2.e119. PMID 12897317
- [Background] Beardslee WR, Salt P, Versage EM, Gladstone TR, Wright EJ, Rothberg PC. Sustained change in parents receiving preventive interventions for families with depression. Am J Psychiatry. 1997 Apr;154(4):510-5. doi: 10.1176/ajp.154.4.510. PMID 9090338
- [Background] Beardslee WR, Wright E, Rothberg PC, Salt P, Versage E. Response of families to two preventive intervention strategies: long-term differences in behavior and attitude change. J Am Acad Child Adolesc Psychiatry. 1996 Jun;35(6):774-82. doi: 10.1097/00004583-199606000-00017. PMID 8682758
- [Background] Betancourt TS, Meyers-Ohki S, Stulac SN, Barrera AE, Mushashi C, Beardslee WR. Nothing can defeat combined hands (Abashize hamwe ntakibananira): protective processes and resilience in Rwandan children and families affected by HIV/AIDS. Soc Sci Med. 2011 Sep;73(5):693-701. doi: 10.1016/j.socscimed.2011.06.053. Epub 2011 Jul 23. PMID 21840634
- [Background] Tol WA, Barbui C, Galappatti A, Silove D, Betancourt TS, Souza R, Golaz A, van Ommeren M. Mental health and psychosocial support in humanitarian settings: linking practice and research. Lancet. 2011 Oct 29;378(9802):1581-91. doi: 10.1016/S0140-6736(11)61094-5. Epub 2011 Oct 16. PMID 22008428
- [Background] Betancourt TS, Borisova II, de la Soudiere M, Williamson J. Sierra Leone's child soldiers: war exposures and mental health problems by gender. J Adolesc Health. 2011 Jul;49(1):21-8. doi: 10.1016/j.jadohealth.2010.09.021. Epub 2010 Dec 24. PMID 21700152
- [Background] Betancourt TS. Attending to the mental health of war-affected children: the need for longitudinal and developmental research perspectives. J Am Acad Child Adolesc Psychiatry. 2011 Apr;50(4):323-5. doi: 10.1016/j.jaac.2011.01.008. No abstract available. PMID 21421171
- [Background] Betancourt TS, Borisova II, Williams TP, Brennan RT, Whitfield TH, de la Soudiere M, Williamson J, Gilman SE. Sierra Leone's former child soldiers: a follow-up study of psychosocial adjustment and community reintegration. Child Dev. 2010 Jul-Aug;81(4):1077-95. doi: 10.1111/j.1467-8624.2010.01455.x. PMID 20636683
- [Background] Betancourt TS, Brennan RT, Rubin-Smith J, Fitzmaurice GM, Gilman SE. Sierra Leone's former child soldiers: a longitudinal study of risk, protective factors, and mental health. J Am Acad Child Adolesc Psychiatry. 2010 Jun;49(6):606-15. doi: 10.1016/j.jaac.2010.03.008. Epub 2010 May 1. PMID 20494270
- [Background] Betancourt TS, Agnew-Blais J, Gilman SE, Williams DR, Ellis BH. Past horrors, present struggles: the role of stigma in the association between war experiences and psychosocial adjustment among former child soldiers in Sierra Leone. Soc Sci Med. 2010 Jan;70(1):17-26. doi: 10.1016/j.socscimed.2009.09.038. Epub 2009 Oct 28. PMID 19875215
- [Background] Betancourt TS, Simmons S, Borisova I, Brewer SE, Iweala U, Soudiere MD. High Hopes, Grim Reality: Reintegration and the Education of Former Child Soldiers in Sierra Leone. Comp Educ Rev. 2008 Nov 1;52(4):565-587. doi: 10.1086/591298. No abstract available. PMID 19337570
- [Background] Betancourt TS, Bass J, Borisova I, Neugebauer R, Speelman L, Onyango G, Bolton P. Assessing local instrument reliability and validity: a field-based example from northern Uganda. Soc Psychiatry Psychiatr Epidemiol. 2009 Aug;44(8):685-92. doi: 10.1007/s00127-008-0475-1. Epub 2009 Jan 22. PMID 19165403
- [Background] Verdeli H, Clougherty K, Onyango G, Lewandowski E, Speelman L, Betancourt TS, Neugebauer R, Stein TR, Bolton P. Group Interpersonal Psychotherapy for depressed youth in IDP camps in Northern Uganda: adaptation and training. Child Adolesc Psychiatr Clin N Am. 2008 Jul;17(3):605-24, ix. doi: 10.1016/j.chc.2008.03.002. PMID 18558315
- [Background] Bolton P, Bass J, Betancourt T, Speelman L, Onyango G, Clougherty KF, Neugebauer R, Murray L, Verdeli H. Interventions for depression symptoms among adolescent survivors of war and displacement in northern Uganda: a randomized controlled trial. JAMA. 2007 Aug 1;298(5):519-27. doi: 10.1001/jama.298.5.519. PMID 17666672
- [Background] Betancourt TS, Speelman L, Onyango G, Bolton P. A qualitative study of mental health problems among children displaced by war in northern Uganda. Transcult Psychiatry. 2009 Jun;46(2):238-56. doi: 10.1177/1363461509105815. PMID 19541749
- [Background] Betancourt TS, Khan KT. The mental health of children affected by armed conflict: protective processes and pathways to resilience. Int Rev Psychiatry. 2008 Jun;20(3):317-28. doi: 10.1080/09540260802090363. PMID 18569183
- [Background] Betancourt TS. Child soldiers: reintegration, pathways to recovery, and reflections from the field. J Dev Behav Pediatr. 2008 Apr;29(2):138-41. doi: 10.1097/DBP.0b013e31816be946. No abstract available. PMID 18408537
- [Background] Betancourt TS, Williams T. Building an evidence base on mental health interventions for children affected by armed conflict. Intervention (Amstelveen). 2008;6(1):39-56. doi: 10.1097/WTF.0b013e3282f761ff. PMID 19997531
- [Background] Betancourt T, Scorza P, Meyers-Ohki S, Mushashi C, Kayiteshonga Y, Binagwaho A, Stulac S, Beardslee WR. Validating the Center for Epidemiological Studies Depression Scale for Children in Rwanda. J Am Acad Child Adolesc Psychiatry. 2012 Dec;51(12):1284-92. doi: 10.1016/j.jaac.2012.09.003. Epub 2012 Nov 8. PMID 23200285
- [Background] Scorza P, Stevenson A, Canino G, Mushashi C, Kanyanganzi F, Munyanah M, Betancourt T. Validation of the "World Health Organization Disability Assessment Schedule for children, WHODAS-Child" in Rwanda. PLoS One. 2013;8(3):e57725. doi: 10.1371/journal.pone.0057725. Epub 2013 Mar 7. PMID 23505437
- [Background] Betancourt TS, Meyers-Ohki SE, Charrow A, Hansen N. Annual Research Review: Mental health and resilience in HIV/AIDS-affected children-- a review of the literature and recommendations for future research. J Child Psychol Psychiatry. 2013 Apr;54(4):423-44. doi: 10.1111/j.1469-7610.2012.02613.x. Epub 2012 Sep 4. PMID 22943414
- [Derived] Betancourt TS, Ng LC, Kirk CM, Brennan RT, Beardslee WR, Stulac S, Mushashi C, Nduwimana E, Mukunzi S, Nyirandagijimana B, Kalisa G, Rwabukwisi CF, Sezibera V. Family-based promotion of mental health in children affected by HIV: a pilot randomized controlled trial. J Child Psychol Psychiatry. 2017 Aug;58(8):922-930. doi: 10.1111/jcpp.12729. Epub 2017 May 15. PMID 28504307